CLINICAL TRIAL: NCT02566096
Title: Efficacy of Transverses Abdominis -Plane Block With Bupivacaine Versus Bupivacaine With Morphine in Patients Undergoing Major Abdominal Cancer Surgery
Brief Title: Efficacy of Transverses Abdominis -Plane Block With Bupivacaine Versus Bupivacaine With Morphine Postoperatively
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 229
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-03

CONDITIONS: Abdominal Cancer
Keywords: major abdominal cancer
MeSH Terms: interventions — Anesthetics, Local; Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP with bupivicaine (Placebo Comparator): 30 patients receive ultrasound guided transversus abdominis-plane block (TAP) with local anesthetic 20 ml of bupivacaine 0.5 % diluted in 20 ml saline (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of the abdominal wall.
  Interventions: Drug: transversus abdominis-plane block with local anesthetic 20 ml of bupivacaine 0.5% + 10 mg morphine
- TAP with bupivicaine with morphine (Active Comparator): 30 patients receive ultrasound guided transversus abdominis-plane block (TAP) with local anesthetic 20 ml of bupivacaine 0.5% + 10 mg morphine diluted in 20 ml saline (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of the abdominal wall.
  Interventions: Drug: transversus abdominis-plane block with local anesthetic 20 ml of bupivacaine 0.5% + 10 mg morphine

INTERVENTIONS:
Drug: transversus abdominis-plane block with local anesthetic 20 ml of bupivacaine 0.5% + 10 mg morphine — compare the analgesic efficacy of transversus abdominis-plane block with bupivicaine with morphine in patients undergoing major abdominal cancer surgery.

SUMMARY:
This study aims to compare the analgesic efficacy of transversus abdominis-plane block with bupivicaine versus bupivacaine with morphine in patients undergoing major abdominal cancer surgery.

DETAILED DESCRIPTION:
This randomized study will be approved by the local ethics committee of South Egypt Cancer Institute, Assuit University, Egypt after written informed consent. This study will include approximately 60 ASA I-II cancer patients with age range (18-60) years, weight (50- 85) kg who will be scheduled for lower abdominal cancer surgery (abdominal hysterectomy, oophorectomy and radical cystectomy). Exclude from the study Patients with known drug allergy to study drugs, significant cardiac, respiratory, renal or hepatic disease, coagulation disorders and those with psychiatric illnesses that would interfere with perception and assessment of pain. Preoperatively, patients will be taught how to evaluate their own pain intensity using the Visual Analog Scale (VAS), scored from 0-10 (where 0= no pain and 10=worst pain imaginable).

Patients will be randomly assigned using an online research randomizer into two groups, 30 patients in each group:

Group 1:

30 patients receive ultrasound guided transversus abdominis-plane block with local anesthetic 20 ml of bupivacaine 0.5 % diluted in 20 ml saline (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of the abdominal wall.

Group 2:

30 patients receive ultrasound guided transversus abdominis-plane block with local anesthetic 20 ml of bupivacaine 0.5% + 10 mg morphine diluted in 20 ml saline (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of the abdominal wall.

Surgery will be performed under standard general anesthesia and ultrasound guided TAP block will be performed before induction of GA.

ELIGIBILITY:
Inclusion Criteria:

* 60 ASA I-II cancer patients with age range (18-60) years,
* weight (50- 85) kg

Exclusion Criteria:

* with patients with known drug allergy to study drugs
* with significant cardiac, respiratory, renal or hepatic disease
* with coagulation disorders
* those with psychiatric illnesses that would interfere with perception and assessment of pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The presence and severity of pain at rest and on coughing will be assessed using a Visual Analog Scale | first 24 hours postoperatively
  The presence and severity of pain at rest and on coughing will be assessed using a Visual Analog Scale will be assessed postoperatively at baseline, 2, 4, 6, 8, 12, 18, and 24 hours.

SECONDARY OUTCOMES:
the level of sedation by using sedation score | 24 hours postoperatively
  the level of sedation by using sedation score (awake and alert = 0, quietly awake = 1, asleep but easily roused= 2, deep sleep = 3) will be assessed postoperatively at baseline, 2, 4, 6, 8, 12, 18, and 24 hours.
first request for analgesia in minutes will be observed | firsr 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Instuite, Asyut, Egypt

REFERENCES:
- [Derived] El Sherif FA, Mohamed SA, Kamal SM. The effect of morphine added to bupivacaine in ultrasound guided transversus abdominis plane (TAP) block for postoperative analgesia following lower abdominal cancer surgery, a randomized controlled study. J Clin Anesth. 2017 Jun;39:4-9. doi: 10.1016/j.jclinane.2017.03.009. Epub 2017 Mar 10. PMID 28494906